CLINICAL TRIAL: NCT06169839
Title: The Effect of Different Simulation Methods Used in Adult Basic Life Support Training on Knowledge, Skills, Self-Efficacy, and Satisfaction in Layperson First Aider
Brief Title: The Effect of Different Simulation Methods Used in Adult Basic Life Support Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Ayşenur YETİK ARAS, Principal Investigator, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AU-N-AYA-01
Record Dates: First submitted 2023-11-24; First posted 2023-12-14 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-06

CONDITIONS: First Aid
Keywords: Adult Basic Life Support; Health Education; Simulation; Layperson First Aider
MeSH Terms: conditions — Health Education

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Skill training with Low Realism Simulation (Active Comparator): the theoretical part of the TYD and OED training with Participation Certificate, the curriculum of which is created by the Ministry of Health, will be explained (by the Researcher). (1 hours) Skill training with Low Realism Simulation (1 hour) Basic CPR Manikin (classical training provided by the Ministry of Health),
  Interventions: Behavioral: Providing BLS and AED trainings given by the Ministry of Health with Low Realism Simulation.
- Skills training with High Reality Simulation (Experimental): the theoretical part of the TYD and OED training with Participation Certificate, the curriculum of which is created by the Ministry of Health, will be explained (by the Researcher). (1 hours) Skills training with High Reality Simulation (1 hour) SimMan® 3G (Laerdal medical)
  Interventions: Behavioral: Providing BLS and AED trainings given by the Ministry of Health with High Reality Simulation
- Skill training will be given with Virtual Reality Application Supported Simulation (Experimental): the theoretical part of the TYD and OED training with Participation Certificate, the curriculum of which is created by the Ministry of Health, will be explained (by the Researcher). (1 hours) Skill training will be given with Virtual Reality Application Supported Simulation (1 hour) and application training will be given with 3D MedSim.
  Interventions: Behavioral: Providing BLS and AED trainings given by the Ministry of Health with Virtual Reality

INTERVENTIONS:
Behavioral: Providing BLS and AED trainings given by the Ministry of Health with Low Realism Simulation. — the theoretical part of the Certificate of Participation TYD and OED training, the curriculum of which is created by the Ministry of Health, will be explained (by the researcher) (1hours). Skill training with Low Realism Simulation (1 hour) Basic CPR Manikin (classical training given by the Ministry of Health),
  Arms: Skill training with Low Realism Simulation
Behavioral: Providing BLS and AED trainings given by the Ministry of Health with High Reality Simulation — the theoretical part of the Certificate of Participation TYD and OED training, the curriculum of which is created by the Ministry of Health, will be explained (by the researcher) (1 hours). Skill training with High Reality Simulation (1 hour) SimMan® 3G (Laerdal medical)
  Arms: Skills training with High Reality Simulation
Behavioral: Providing BLS and AED trainings given by the Ministry of Health with Virtual Reality — the theoretical part of the Certificate of Participation TYD and OED training, the curriculum of which is created by the Ministry of Health, will be explained (by the researcher) (1 hours). Skill training with Virtual Reality Application Supported Simulation (1 hour) Application training will be given with 3D MedSim.
  Arms: Skill training will be given with Virtual Reality Application Supported Simulation

SUMMARY:
The aim of this study is to evaluate the effects of different simulation methods Virtual Reality-Aided Simulation (VRS), High-Fidelity Simulation (HFS), Low-Fidelity Simulation (LFS) used in adult Basic Life Support (BLS) training on the knowledge, skills, self-efficacy, and satisfaction levels of lay rescuers who are not health professionals.

DETAILED DESCRIPTION:
The study population included Ministry of Health personnel, and the sample comprised participants of the certified BLS training held on December 3-6, 2023. Sample size was calculated using G*Power (v3.1.9), based on a medium effect size (f = 0.25), with α = 0.05, power = 0.90, three groups, and two time points. The analysis indicated a minimum of 54 participants; accounting for possible dropouts, 21 individuals were included per group, totaling 63 volunteers. The data collection instruments included the Descriptive Characteristics Form, the General Self-Efficacy Scale (GSES), the BLS Knowledge Level Assessment Form, the BLS Skills Evaluation Form, the BLS Self-Efficacy Questionnaire, and the BLS Training Satisfaction Survey.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily agreeing to participate in the research
* Being between the ages of 18-65
* Having applied for Basic life support and Automatic external defibrillator training with a participation certificate issued by the Ministry of Health.
* Being a Ministry of Health personnel.

Exclusion Criteria:

* Refusal to participate in the research
* Becoming a health professional
* Receiving previously authorized basic first aid training.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2023-12-06 (Actual); Primary Completion 2024-03-08 (Actual); Study Completion 2025-06-29 (Actual)

PRIMARY OUTCOMES:
Basic Life Support (BLS) Knowledge Level Evaluation | 3 months
  20 multiple-choice questionnaires aimed at measuring the BLS knowledge level prepared by the researcher in line with the relevant literature. It is evaluated on the basis of the highest 20 and the lowest 0 points. Getting high scores from the questions indicates a high level of BLS knowledge. Application process; pre-test, post-training post-test and 3-month post-test.
Basic Life Support Application Skill | 3 months
  Basic Life Support Application Skill Form and CPR effectiveness : BLS skill evaluation form used by the Ministry of Health. It consists of 11 questions. The highest score is 20 and the lowest is 0. Getting high scores from the questions indicates a high level of BLS skill level. CPR effectiveness (compression rate, depth and chest recoil) will be measured via a QCPR manikin.
  Application process; post-training test and 3-month post-test.
Basic Life Support Self-Efficacy | 3 months
  It was created to measure self-efficacy in emergency CPR, based on the General Self-Efficacy Scale. 4 items are 7-point Likert type. Getting high scores on the items indicates a high level of general self-efficacy. Application process; post-training test and 3-month post-test.
Basic Life Support Training Satisfaction | 3 days
  A choice will be made between 0 and 10. "0" indicates I am not satisfied at all, "10" indicates I am very satisfied. Application process; post-training testing.

SECONDARY OUTCOMES:
General Self-Efficacy Scale (GÖYS) | 3 days
  The number of items is 10. The scale was prepared as a 4-point Likert type. Getting high scores on the items indicates a high level of general self-efficacy. Application process; pre-training test.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Ankara University, Nursing Faculty, Ankara, Altindağ
  - T.R. Ministry of Health Bilkent Campus Universiteler District Şehit Mehmet Bayraktar Caddesi, Ankara

IPD SHARING:
Plan to Share IPD: Undecided